CLINICAL TRIAL: NCT06857617
Title: A Phase 1/2 Randomized Placebo-Controlled Double-Blind Study to Investigate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Doses of MET097 in Adult Participants With Obesity and Overweight But Otherwise Healthy
Brief Title: This Study Will Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of MET097 in Adult Participants With Overweight or Obesity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Metsera, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MET097-23-101
Record Dates: First submitted 2025-01-14; First posted 2025-03-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Part A (72 participants), Part B (70 participants), Part C (120 participants)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- (Part C) MET097 (Experimental): Once-weekly subcutaneous injection of MET097 for 13 weeks
  Interventions: Biological: (Part C) MET097
- (Part C) Placebo (Placebo Comparator): Once-weekly subcutaneous injection of Placebo for 13 weeks
  Interventions: Biological: (Part C) Placebo

INTERVENTIONS:
Biological: (Part C) MET097 — Participants will receive 13 once-weekly subcutaneous injections of MET097 as follows:
  * 12 once-weekly doses of 0.6mg followed by a 13th dose of 1.2mg
  * 12 once-weekly doses of 0.6mg followed by a 13th dose of 2.4 mg
  * 12 once-weekly doses of 0.8 mg followed by a 13th dose of 1.6 mg
  * 12 once-weekly doses of 0.8 mg followed by a 13th dose of 3.2 mg
  * 12 once-weekly doses of 1.0 mg followed by a 13th dose of 2.0 mg
  * 12 once-weekly doses of 1.0 mg followed by a 13th dose of 4.0 mg
  * 12 once-weekly doses of 1.2 mg followed by a 13th dose of 2.4 mg
  * 12 once-weekly doses of 1.2 mg followed by a 13th dose of 4.8 mg
  * Titration regimen of 0.4mg/0.8mg/1.2mg with 4 doses at each dose-level, followed by a 13th dose of 2.4mg
  * Titration regimen of 0.4mg/0.8mg/1.2mg with 4 doses at each dose-level, followed by a 13th dose of 4.8mg
  Arms: (Part C) MET097
Biological: (Part C) Placebo — Participants will receive 13 once-weekly subcutaneous injections of matching placebo
  Arms: (Part C) Placebo

SUMMARY:
The goal of this Phase 1/2 clinical trial is to assess the safety, tolerability, pharmacokinetics, and efficacy of once-weekly subcutaneous injections of MET097 in otherwise healthy adults with overweight or obesity.

The trial will be conducted in three parts. Part A consists of single ascending dose (SAD) cohorts of MET097 or placebo. Part B consists of multiple ascending dose (MAD) cohorts, with participants treated with five once-weekly doses of MET097 or placebo. In Part C, participants will receive once-weekly doses of MET097 or placebo for 12 weeks, followed by a single dose at 2X or 4X to explore the potential for once-monthly dosing.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/Obese but otherwise healthy adult male or female with a BMI within 27.0 kg/m2 to 38.0 kg/m2, inclusively
* At least 18 years of age but not older than 70 years of age
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an Investigator
* Estimated glomerular filtration rate (eGFR) ≥90 mL/min at the Screening visit

Exclusion Criteria:

* Female who is lactating or who is pregnant according to the pregnancy test at the Screening visit or prior to the first study drug administration
* Seated blood pressure higher than 160/95 mmHg at the Screening visit
* Elevated resting pulse greater than 100 beats per minute at Screening visit
* Presence of clinically significant ECG abnormalities
* Diagnosis of diabetes (type 1 or type 2)
* Participation in a weight loss program with or without pharmacotherapy during the 3 months prior to study administration
* Obesity induced by endocrinologic disorders (e.g., Cushing's syndrome) or diagnosed monogenetic or syndromic forms of obesity (e.g., Melanocortin 4 Receptor deficiency or Prader-Willi Syndrome).
* Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia type

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
(Part C) Percent change from baseline in body weight at Week 12 (Day 85). | Day 1 (Week 0) to Day 85 (Week 12)

SECONDARY OUTCOMES:
(Part C) To characterize the maximum observed concentration (Cmax). | Day 1 (Week 0) to Day 160 (Week 31)
(Part C) To characterize the time of maximum observed concentration (Tmax). | Day 1 (Week 0) to Day 160 (Week 31)
(Part C) To characterize the area under the concentration versus time curve (AUC). | Day 1 (Week 0) to Day 160 (Week 31)
(Part C) To characterize the elimination half-life (t1/2). | Day 1 (Week 0) to Day 160 (Week 31)
(Part C) Occurrence of treatment-emergent adverse events (TEAEs) through Week 12. | Day 1 (Week 0) to Day 85 (Week 12)
(Part C) Occurrence of TEAEs following the 13th dose. | Day 85 (Week 12) to Day 160 (Week 31)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site MET097 23-101-002, Anaheim, California
  - Research Site MET097 23-101-003, Cypress, California
  - Research Site MET097 23-101-001, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: Undecided